CLINICAL TRIAL: NCT01066507
Title: Concordance Study for Amplification Detection of Her2 FISH in Breast Tissue Sections
Brief Title: Detection of Amplification of Her2 Fluorescent in Situ Hybridization (FISH) in Breast Tissue Sections
Acronym: Her2F test
Status: Completed | Type: Observational
Sponsor: Applied Spectral Imaging Ltd. (Industry)
Responsible Party: Tsafrir Kolatt, Applied Spectral Imaging Ltd.
Other Study IDs: ASI-Her2F
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Breast Cancer
Keywords: Her2; FISH; Breast cancer; Amplification
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Paraffin embedded tissue sections
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer: Slides containing breast cancer paraffin embedded tissue sections.

SUMMARY:
The purpose of the study is the identification of amplification level in human breast tissue. The imaging system is intended for diagnostic use as an aid to the pathologist in the detection, counting and classification of Her2 FISH stained tissue samples.

ELIGIBILITY:
Inclusion Criteria:

* Well stained breast tissue slides with bright Her2 signals

Exclusion Criteria:

* Very old slides that were already bleached

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The breast samples were taken from female patients after cut biopsies. Paraffin embedded blocks were prepared and the secssion slides were stained with the PathVysion prove for Her2 FISH applification detection
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Dobin, Ph.D., Study Director — Section Chief, Cytogenetics
Locations (3):
- United States (2):
  - PLUS Diagnostics, Lakewood, New Jersey
  - Scott & White Hospital, Texas, Temple, Texas
- Sheba Medical Center, Pathology Dep., Tel Aviv, Israel